CLINICAL TRIAL: NCT01666522
Title: Effect of Vitamin D Supplementation and Physical Activity in Preventing Sarcopenia in Older Adults With Osteoporosis
Brief Title: Vitamin D and Physical Activity for Prevention of Sarcopenia in Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: alexmed116671002
Record Dates: First submitted 2012-08-03; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Sarcopenia
Keywords: sarcopenia; osteopenia/osteoporosis; older adults; vitamin D supplementation; physical activity
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic; Motor Activity | interventions — Vitamin D; Cholecalciferol; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D (Experimental): vitamin D-oral cholecalciferol 2000 IU/day for 4 months
  Interventions: Drug: Vitamin D
- Physical activity (Active Comparator): A 3-day/week exercise programme lasting 60 minutes each day for 4 months was instigated.
  Interventions: Other: Physical activity
- Vitamin D and Physical activity (Experimental): Vitamin D -oral cholecalciferol 2000 IU/day and Physical activity-60-minute 3-day/week exercise programme
  Interventions: Drug: Vitamin D; Other: Physical activity
- Control (Placebo Comparator): The control group was provided with health education using videotaped presentations, physician talks on topics concerning bone and muscle health.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — vitamin D given orally as tablets at a dosage of 2000 IU/day for 4 months
  Other Names: cholecalciferol
  Arms: Control; Vitamin D; Vitamin D and Physical activity
Other: Physical activity — Physical activity in the form of an exercise programme consisting of 60 minutes all inclusive warming up , strengthening, resistance and stretching exercises were instigated 3 times a week for 4 months.
  Other Names: Exercise programme
  Arms: Physical activity; Vitamin D and Physical activity

SUMMARY:
In the present study the aim was to determine the prevalence of sarcopenia and to evaluate the effectiveness of an exercise program and vitamin D supplementation in enhancing muscle mass and strength in community-dwelling older adults with osteopenia /osteoporosis.

One hundred and forty-five individuals aged 65 years and above with documented osteopenia/osteoporosis were scanned for sarcopenia. The participants were randomly assigned to one of four groups: Group 1-PA and vitamin D (n= 38), Group 2-PA(n=36), Group 3-vitamin D (n= 36) or Group 4-healthy lifestyle(n =35) for 16 weeks. The PA group received a 60-minute 3-day/week exercise programme, the vitamin D group received oral cholecalciferol 2000 IU/day and the control group was provided with health education using videotaped presentations, physician talks on topics concerning bone and muscle health. Body composition was measured DEXA. Vitamin D levels were measured and PA was measured using the Baecke Physical Activity Questionnaire. Physical performance was assessed using upper limb grip strength, walking speed and knee extension strength. All data was collected at baseline and at 4 months.

DETAILED DESCRIPTION:
Ageing is associated with changes in body composition and due to the ageing of the populations and the lessened physical activity (PA), sarcopenia and osteopenia /osteoporosis are emerging as major health concerns. Lack of PA is a significant risk factor for sarcopenia. Vitamin D plays an important role on bone and muscle development.

This study was conducted to determine the prevalence of sarcopenia and to evaluate the effectiveness of PA and vitamin D supplementation in enhancing muscle mass and strength in community-dwelling older adults with osteopenia /osteoporosis.\ One hundred and forty-five individuals aged 65 years and above with documented osteopenia/osteoporosis were scanned for sarcopenia (defined as a relative skeletal muscle index (appendicular skeletal muscle mass divided by height) below 5.45 kg/m2). The participants were randomly assigned to one of four groups: Group 1-PA and vitamin D (n= 38), Group 2-PA(n=36), Group 3-vitamin D (n= 36) or Group 4-healthy lifestyle(n =35) for 16 weeks. The PA group received a 60-minute 3-day/week exercise programme, the vitamin D group received oral cholecalciferol 2000 IU/day and the control group was provided with health education using videotaped presentations, physician talks on topics concerning bone and muscle health. Body composition was measured by dual energy X-ray absorptiometry (DEXA). Vitamin D levels were measured by Liaison immunoassay. PA was measured using the Baecke Physical Activity Questionnaire. Physical performance was assessed using upper limb grip strength, walking speed and knee extension strength. All data was collected at baseline and at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 60 and above
* osteopenia/osteoporosis

Exclusion Criteria:

* severe cognitive impairment
* major organ disease
* current consumption of corticosteroids or vitamin D

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
muscle mass change | 4 months
Muscle mass change | 4 months
  To determine change in vitamin D status, fasting blood samples were collected from all participants at baseline and after 16 weeks of intervention and were measured by Liaison immunoassay.
  Muscle mass change and sarcopenia prevention was measured using the relative skeletal muscle index (appendicular skeletal muscle mass divided by height) below 5.45 kg/m2).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Alexandria Governorate, Egypt